CLINICAL TRIAL: NCT02860286
Title: A Multicenter Study of the EZH2 Inhibitor Tazemetostat in Adult Subjects With Relapsed or Refractory Malignant Mesothelioma With BAP1 Loss of Function
Brief Title: Study of the EZH2 Inhibitor Tazemetostat in Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-203
Record Dates: First submitted 2016-07-27; First posted 2016-08-09 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Mesothelioma; BAP1 Loss of Function
MeSH Terms: conditions — Mesothelioma | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Tazemetostat (Experimental): Oral Tazemetostat 800mg BID
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2 gene.
  Other Names: EPZ-6438; E7438

SUMMARY:
This is a Phase 2, multicenter, open-label, 2-part, single-arm, 2-stage study of tazemetostat 800 mg two times a day (BID) administered orally. Screening of subjects to determine eligibility for the study will be performed within 21 days of the first planned dose of tazemetostat.

In Part 1: planned to enroll 12 subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status will be treated and undergo pharmacokinetics (PK) blood sample collection after a single tazemetostat 800 mg.

Part 2 plans to include 55 subjects with BAP1-deficient relapsed or refractory malignant mesothelioma.

Treatment with tazemetostat will continue until disease progression, unacceptable toxicity or withdrawal of consent, or termination of the study. Response assessment will be evaluated after 6 weeks of treatment and then every 12 weeks thereafter while on study.

ELIGIBILITY:
Inclusion Criteria:

1. Age (at the time of consent) ≥18 years of age
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Has a life expectancy of >3 months
4. Has mesothelioma (pleural, peritoneal, pericardial, tunica vaginalis) of any histology that is relapsed or refractory after treatment with at least one pemetrexed-containing regimen
5. Has a documented local diagnostic pathology of original biopsy confirmed by a Clinical Laboratory Improvement Amendments (CLIA)/College of American Pathologists (CAP) or equivalent laboratory certification
6. Part 2: Molecular evidence of BAP1 loss of function mutation present on local pathology, e.g., lack of nuclear BAP1 staining by immunohistochemistry (IHC) or evidence of loss of function by gene sequencing
7. Has sufficient archival tumor tissue (a minimum of 10 slides or tumor block) available for central retrospective testing of BAP1 status
8. Has all prior treatment (i.e., chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤ Grade 1 per CTCAE, version 4.03 or are clinically stable and not clinically significant, at time of enrollment
9. Prior therapy(ies), if applicable, must be completed according to the criteria below prior to first dose of tazemetostat:

   * Cytotoxic chemotherapy; at least 21 days since last dose
   * Non-cytotoxic chemotherapy (e.g., small molecule inhibitor); at least 14 days since last dose
   * Monoclonal antibody; at least three half-lives since the last dose
   * Non-antibody immunotherapy (e.g., tumor vaccine); at least 42 days since last dose
   * Radiotherapy, at least 14 days from last local site radiotherapy
   * Hematopoietic growth factor; at least 14 days from last dose
   * Investigational drug; 30 days or five half-lives, whichever is longer, from last dose
10. Has measurable disease based on either modified RECIST [Nowak 2005] for thoracic disease or RECIST 1.1 elsewhere
11. Has adequate hematologic (bone marrow and coagulation factors), renal, and hepatic function as defined by criteria below:

    * Hemoglobin ≥9 mg/dL
    * Platelets ≥100,000/mm3 (≥100 × 109/L) without platelet transfusion for 7 days
    * ANC ≥1000/mm3 (≥1.0 × 109/L) without growth factor support for 14 days
    * Coagulation: Prothrombin time (PT) <1.5 × ULN and partial thromboplastin time (PTT) <1.5 × ULN
    * Creatinine < 2.0 × ULN
    * Hepatic function: Conjugated bilirubin <1.5 × ULN and ALT and AST <3 × ULN
12. Has a QT interval corrected by Fridericia's formula (QTcF) ≤480 msec
13. Willing to provide tissue for translational research
14. Female subjects of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study drug; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required and subject also should agree to use an adequate method of contraception starting with screening through 30 days after the last dose of study therapy (if sexually active).
15. Male subjects should agree to use condoms starting with the first dose of study therapy through 30 days after the last dose of study therapy if sexually active with a female of childbearing potential

Exclusion Criteria:

1. Has had prior exposure to tazemetostat or other inhibitor(s) of enhancer of zeste homologue-2 (EZH2)
2. Has a history of known central nervous system metastasis
3. Has had a prior malignancy other than the malignancies under study Exception: A subject who has been disease-free for 5 years, or a subject with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is eligible.
4. Has had major surgery within 3 weeks prior to enrollment (a percutaneous biopsy, pleural catheter insertion, placement of central venous catheter or other minor procedure are permitted)
5. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from time of enrollment throughout their time on study
6. Has cardiovascular impairment, history of congestive heart failure greater than NYHA Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months prior to the planned first dose of tazemetostat; or ventricular cardiac arrhythmia requiring medical treatment
7. Is currently taking any prohibited medication(s)
8. Has an active infection requiring systemic treatment
9. Has a congenital or acquired immunodeficiency, including subjects with known history of infection with human immunodeficiency virus (HIV) NOTE: HIV-positive subjects who are taking antiretroviral therapy are ineligible due to potential PK interactions with tazemetostat.
10. Has known history of chronic infection with hepatitis B virus (hepatitis B surface antigen positive) or hepatitis C virus (detectable anti-hepatitis C circulating viral RNA)
11. Has had a deep venous thrombosis (DVT) or pulmonary embolism within the 3 months prior to study enrollment.

    NOTE: Subjects with a history of a DVT or pulmonary embolism >3 months prior to study enrollment who are on anticoagulation therapy with low molecular weight heparin are eligible for this study.
12. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - City of Hope National Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
- France (3):
  - Institut Bergonie, Bordeaux
  - CHRU de Lille, Lille
  - Institut Gustave Roussy, Villejuif
- United Kingdom (6):
  - University of Leicester & Leicester University Hospitals, Leicester
  - St. Bartholomew's Hospital, London
  - University College Hospital, London
  - Royal Marsden Hospital - Chelsea, London
  - University Hospital of South Manchester, Manchester
  - Royal Marsden Hospital - Surrey, Sutton

IPD SHARING:
Plan to Share IPD: No
To be determined.

REFERENCES:
- [Derived] Zauderer MG, Szlosarek PW, Le Moulec S, Popat S, Taylor P, Planchard D, Scherpereel A, Koczywas M, Forster M, Cameron RB, Peikert T, Argon EK, Michaud NR, Szanto A, Yang J, Chen Y, Kansra V, Agarwal S, Fennell DA. EZH2 inhibitor tazemetostat in patients with relapsed or refractory, BAP1-inactivated malignant pleural mesothelioma: a multicentre, open-label, phase 2 study. Lancet Oncol. 2022 Jun;23(6):758-767. doi: 10.1016/S1470-2045(22)00277-7. Epub 2022 May 16. PMID 35588752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study EZH-203 was conducted at 16 clinical sites in France, UK, and USA. Subjects were screened for eligibility within 21 days of the planned date of the first dose of tazemetostat.
  Eligible subjects were enrolled into 2 different parts:
  * Part 1 - Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status
  * Part 2 - Subjects with relapsed or refractory BAP1-deficient malignant mesothelioma.
Pre-assignment Details: Seventy-four subjects were enrolled and treated with study drug (13 subjects in Part 1 and 61 subjects in Part 2).
  No patients were excluded due to unmet study eligibility criteria.
Groups:
- Part 1 (Pharmacokinetics): Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status were to be treated and PK blood samples collected after a single tazemetostat 800 mg dose on Cycle 1 Day 1 and after repeated twice daily doses of tazemetostat 800 mg on Cycle 1 Day 15. Subjects were to receive a single oral 800 mg tazemetostat dose on Cycle 1 Day 1. Starting on Cycle 1 Day 2, tazemetostat was orally administered at a dose of 800 mg twice daily.
- Part 2 (Efficacy): subjects with BAP1-deficient relapsed or refractory malignant mesothelioma were to receive orally administered tazemetostat 800 mg twice daily starting on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Part 1 (Pharmacokinetics) | Part 2 (Efficacy)
Started | 13 | 61
Completed | 13 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 (Pharmacokenitc): Subjects enrolled in Part 1were to receive a single 800 mg tazemetostat dose on Cycle 1 Day 1. Starting on Cycle 1 Day 2, tazemetostat was to be administered at a dose of 800 mg twice daily. PK blood samples were to be collected after administration of a single dose of 800 mg tazemetostat on Cycle 1 Day 1 and after repeated twice daily doses of tazemetostat 800 mg on Cycle 1 Day 15. Plasma samples were to be analyzed for tazemetostat after each set of 6 subjects completed the PK sampling procedures on Cycle 1 Day 15.
- Part 2 (Efficacy): In Part 2, subjects with BAP1-deficient relapsed or refractory malignant mesothelioma were to receive orally administered tazemetostat 800 mg twice daily starting on Cycle 1 Day 1.
  A 2-stage Green-Dahlberg design was utilized with a stopping rule to allow early termination at the end of Stage 1 if there was strong evidence of lack of efficacy based on results from the first 30 treated subjects who completed at least the 12-week assessment, completed the final study visit, or terminated early from the study, whichever was sooner. If early stopping criteria were met, enrollment was to be stopped. To avoid disruptions in the study, enrollment and treatment of subjects were not halted in order to conduct the interim analysis.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Pharmacokenitc) | Part 2 (Efficacy) | Total
Number analyzed (Participants) | 13 | 61 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 37 | 43
  >=65 years | 7 | 24 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (8.58) | 65.1 (10.56) | 65.0 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 22 | 25
  Male | 10 | 39 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 44 | 49
  Other | 6 | 15 | 21
Region of Enrollment [Number; unit: participants]
  United States | 8 | 15 | 23
  United Kingdom | 2 | 35 | 37
  France | 3 | 11 | 14
Baseline Disease Characteristics and Prior Therapies [Count of Participants; unit: Participants]
  Solid Tumor with 1 prior line of systemic Anticancer Therapy | 3 | 27 | 30
  Solid Tumor with 2 prior lines of systemic Anticancer Therapy | 7 | 13 | 20
  Solid Tumor with 3 prior lines of systemic Anticancer Therapy | 1 | 14 | 15
  Solid Tumor with 4 prior lines of systemic Anticancer Therapy | 1 | 1 | 2
  Solid Tumor with >=5 prior lines of systemic Anticancer Therapy | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacokinetics Profile of Tazemetostat and Its Metabolite (Plasma): Cmax
Description: To assess the pharmacokinetic (PK) and safety profile of single (Cycle 1 day 1) and repeated doses (Cycle 1 day 2 onwards) of 800 mg tazemetostat administered as 400 mg tablets in subjects with relapsed or refractory malignant mesothelioma regardless of BRCA1 associated protein 1 (BAP1) status.
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 12 post-dose
Measure: Mean (Standard Deviation); unit: Ng/mL
Groups:
- Part 1 (Pharmacokinetics): Assessment of pharmacokinetic (PK) and safety profile of single (Cycle 1 day 1) and repeated doses (Cycle 1 day 2 onwards) of 800 mg tazemetostat administered as 400 mg tablets in subjects with relapsed or refractory malignant mesothelioma regardless of BRCA1 associated protein 1 (BAP1) status.
Arm/Group | Part 1 (Pharmacokinetics)
Number analyzed (Participants) | 13
Ng/mL | 933 (440)

2. Primary Outcome: Part 1: Pharmacokinetics Profile of Tazemetostat and Its Metabolite (Plasma): Tmax
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and12 post-dose.
Measure: Median (Inter-Quartile Range); unit: Hour
Arm/Group | Part 1 (Pharmacokinetics)
Number analyzed (Participants) | 13
Hour | 1.1 [1 to 4]

3. Primary Outcome: Part 1: Pharmacokinetics Profile of Tazemetostat and Its Metabolite (Plasma): AUC(0-t)
Description: as for outcome 1
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and12 post-dose.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (Pharmacokinetics)
Number analyzed (Participants) | 13
h*ng/mL | 3650 (1640)

4. Primary Outcome: Part 1: Pharmacokinetics Profile of Tazemetostat and Its Metabolite (Plasma): AUC(0-∞)
Description: Pharmacokinetics profile of tazemetostat and its metabolite (plasma) assessing AUC(0-∞)
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 12 post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (Pharmacokinetics)
Number analyzed (Participants) | 13
h*ng/mL | 3410 (1640)

5. Primary Outcome: Part 1: Pharmacokinetics Profile of Tazemetostat and Its Metabolite (Plasma): t1/2
Description: Results from assessing the half-life of Tazemetostat and its metabolite shown below
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 12 post-dose
Measure: Mean (Standard Deviation); unit: Hour
Groups:
- Part 1(Pharmacokinetics): Oral Tazemetostat 800mg BID
  Tazemetostat: Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2 gene.
Arm/Group | Part 1(Pharmacokinetics)
Number analyzed (Participants) | 13
Hour | 3.06 (0.307)

6. Primary Outcome: Part 2: To Assess Disease Control Rate (DCR) Defined as Number of Subjects With Complete Response (CR), Partial Response (PR) and Stable Disease (SD)
Description: Overall, the disease control rate (DCR) (calculated as subjects with CR + subjects with PR + subjects with SD at 12 weeks in duration), and the DCR at 24 weeks.
Time Frame: The patients were assessed for DCR for up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Subjects with relapsed or refractory BAP1-deficient malignant mesothelioma.
Arm/Group | Part 2
Number analyzed (Participants) | 61
Participants
  DCR at 12 weeks | 33
  DCR at 24 weeks | 20

7. Primary Outcome: Incidence of Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Time Frame: From the first dose of study treatment until the earlier of either 30 days after the discontinuation of study treatment or until the initiation of subsequent anticancer therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Subjects with relapsed orrefractory malignantmesothelioma regardless ofBAP1 status were to be treatedand PK blood samplescollected after a singletazemetostat 800 mg dose onCycle 1 Day 1 and afterrepeated twice daily doses oftazemetostat 800 mg on Cycle1 Day 15. Subjects were toreceive a single oral 800 mgtazemetostat dose on Cycle 1Day 1. Starting on Cycle 1 Day2, tazemetostat was orallyadministered at a dose of 800mg twice daily.
- Part 2: Subjects with BAP1-deficientrelapsed or refractorymalignant mesothelioma wereto receive orally administeredtazemetostat 800 mg twicedaily starting on Cycle 1 Day1
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 13 | 61
Participants
  Any TEAE | 13 | 60
  Any TEAE Grade 3 or 4 | 5 | 31
  Any Treatment-Related TEAE | 8 | 44
  Any Treatment-Related TEAE Grade 3 or 4 | 3 | 9
  Any TEAE Leading to Dose Reduction or 4or() { | 0 | 3
  Any TEAE Leading to Study Drug Interruption�� | 5 | 22
  Any TEAE Leading to Study Drug Discontinuation | 0 | 2
  Any TESAENR | 2 | 23
  Any Treatment-Related TESAE | 1 | 2
  Any Protocol Defined AE of Special Interestion | 0 | 0

8. Secondary Outcome: Part 1 and 2: Objective Response Rate (ORR; Complete Response + Partial Response [CR + PR])
Description: ORR (confirmed CR+PR) to tazemetostat in subjects with relapsed/refractory malignant mesothelioma using disease-appropriate standardized response criteria (modified RECIST or RECIST 1.1)
Time Frame: Assessed every 6 weeks for duration of study participation which is estimated to be 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 13 | 61
Participants
  Objective Response Rate, | 0 | 2
  Complete response | 0 | 0
  Partial response | 0 | 2

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-Free Survival is defined as the interval of time between the date of the first dose of study drug and the earliest date of disease progression or death due to any cause. PFS was analyzed and listed for the ITT population. PFS was calculated using the Kaplan-Meier method.
Time Frame: The patients were assessed for PFS for up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Part 1: Part 1 - Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status
  Part 2: Subjects with relapsed or refractory BAP1-deficient malignant mesothelioma
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 13 | 61
Weeks | 12 [5.4 to 34.1] | 18 [1.6 to 114.3]

10. Secondary Outcome: Part 1 and 2: Overall Survival (OS)
Description: OS was analyzed and listed for the ITT population. Subjects who have not died were censored at the date of last contact which was identified from a visit date, study assessment (physical examination, vital signs, ECOG performance status, electrocardiogram [ECG], study drug record, radiological evaluation), AE, medication, or disposition information.
  OS was calculated using the Kaplan-Meier method. OS at 12 and 24 weeks along with the associated 2-sided 95% CIs were provided. Median OS, first and third quartiles and associated 95% 2-sided CIs were provided.
Time Frame: The patients were assessed for PFS for up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 13 | 61
Weeks | 29.0 [16.3 to 139.7] | 41.0 [1.6 to 120.9]

11. Secondary Outcome: Part 1 and 2: To Evaluate the Duration of Response (DOR) in Subjects With Confirmed CR or PR
Description: DOR was calculated for subjects with a confirmed CR or PR. DOR is defined as the time from the date of the initial response (CR/PR) to the date of first documented PD or death due to any cause, whichever occurs first.
  DOR censoring rules followed those of the PFS analysis defined in the SAP. DOR was analyzed using the Kaplan-Meier methods and the median DOR, first quartile, and third quartile was presented. The associated 2- sided 95% CIs was estimated.
Time Frame: Every 6 weeks up to disease progression or start of new anti-cancer therapy assessed for up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 statu
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 13 | 61
Participants
  DOR great than 6 weeks | 0 | 0
  DOR great than 12 weeks | 0 | 0
  DOR great than 18 weeks | 0 | 2

12. Secondary Outcome: Part 1: To Assess Disease Control Rate (DCR) Defined as Number of Subjects With Complete Response (CR), Partial Response (PR) and Stable Disease (SD)
Description: as for outcome 6
Time Frame: The patients were assessed for DCR for up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Part: Subjects with relapsed or refractory malignant mesothelioma regardless of BAP1 status
Arm/Group | Part
Number analyzed (Participants) | 13
Participants
  DCR at 12 weeks | 5
  DCR at 24 weeks | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a period of 2 years.
Description: No other adverse events are listed in the CSR.
Groups:
- Part 1 (Pharmacokinetics): Assessed the pharmacokinetic (PK) and safety profile of single (Cycle 1 day 1) and repeated doses (Cycle 1 day 2 onwards) of 800 mg tazemetostat administered as 400 mg tablets in subjects with relapsed or refractory malignant mesothelioma regardless of BRCA1 associated protein 1 (BAP1) status.
- Part 2 (Efficacy): To assess disease control rate (DCR) at 12 weeks (consisting of complete response [CR], partial response [PR], or stable disease [SD]) according to modified RECIST (Nowak, 2005) for thoracic disease or RECIST 1.1 elsewhere in subjects with relapsed or refractory BAP1-deficient malignant mesothelioma treated with tazemetostat
Arm/Group | Part 1 (Pharmacokinetics) | Part 2 (Efficacy)
All-Cause Mortality (participants affected / at risk) | 1/13 | 7/61
Serious Adverse Events (participants affected / at risk) | 2/13 | 4/61
Other Adverse Events (participants affected / at risk) | 13/13 | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Pharmacokinetics) (N=13) | Part 2 (Efficacy) (N=61)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Air embolism (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave inversiontion (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Pharmacokinetics) (N=13) | Part 2 (Efficacy) (N=61)
Nausea (Gastrointestinal disorders) | 6 (6) | 15 (22)
Vomiting (Gastrointestinal disorders) | 2 (4) | 15 (18)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 5 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 22 (28)
Asthenia (General disorders) | 1 (1) | 8 (10)
Oedema peripheral (General disorders) | 1 (1) | 6 (8)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Chills (General disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (13) | 14 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 17 (17)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Irritation (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 8 (11)
Upper respiratory Tract Infection (Infections and infestations) | 1 (1) | 5 (5)
Oral candidiasis (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 22 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 18 (33)
Dysgeusia (Nervous system disorders) | 0 (0) | 8 (11)
Dizziness (Nervous system disorders) | 0 (0) | 4 (5)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 12 (15)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 13 (17)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02860286/Prot_SAP_000.pdf